CLINICAL TRIAL: NCT02575703
Title: Disposition of [¹⁴C]-LY3023414 Following Oral Administration in Healthy Subjects
Brief Title: A Study of [¹⁴C]-LY3023414 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15697; I6A-EW-CBBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-10-05; First posted 2015-10-15 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — LY3023414

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [¹⁴C]-LY3023414 (Experimental): Single oral dose of [¹⁴C]-LY3023414 administered on Day 1
  Interventions: Drug: [¹⁴C]-LY3023414

INTERVENTIONS:
Drug: [¹⁴C]-LY3023414 — LY3023414 in solution containing approximately 100 microCi [¹⁴C]-LY3023414

SUMMARY:
This type of study is called a radiolabeled study. For this study, LY3023414 has been specially prepared to contain the radioactive carbon atom [¹⁴C]. [¹⁴C] is a naturally occurring radioactive form of the element carbon. Adding a low dose of radiation to the study drug does not change how the drug works but helps to identify when the drug appears in the blood, urine, breath, and stool after it is given. The study will last about 15 days for each participant, not including screening. Screening is required within 28 days prior to enrollment. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women

  * Male participants: Will be sterile (including vasectomy), confirmed by documentation. Men who are sexually active with a pregnant partner agree to use a condom for 91 days from the time of dosing
  * Female participants: Women not of childbearing potential due to surgical sterilization (at least 6 months after hysterectomy with or without bilateral oophorectomy or at least 6 months after tubal ligation) confirmed by medical history or menopause. Postmenopausal women include women with spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (eg, oral contraceptives, hormones, gonadotropin releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy) and a follicle-stimulating hormone level greater than 40 milli international units per milliliter (mIU/mL)
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per meter square (kg/m²)
* Have clinical laboratory test results within normal reference range for the population or investigator site
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Have participated in a [¹⁴C]-study within the last 6 months prior to admission for this study. The total 12-month exposure from this study and a maximum of one other previous [¹⁴C]-study within 6 to 12 months of this study must be within the Code of Federal Regulations (CFR) recommended levels considered safe: Less than 5000 millirem (mrem)/year whole body exposure.
* Exposure to significant diagnostic, therapeutic, or employment-related radiation within 12 months prior to dosing (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Are participants who have previously completed or withdrawn from this study or any other study investigating LY3023414, and have previously received the investigational product
* Have known allergies to LY3023414, related compounds, or any components of the formulation
* Regularly use known drugs of abuse and/or show positive findings on urinary drug testing
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Intend to use over-the-counter or prescription medication within 7 days prior to dosing
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week, or are unwilling to stop alcohol consumption from 48 hours prior to admission and while resident in the Clinical Research Unit (CRU)
* Have consumed herbal supplements, grapefruits or grapefruit-containing products, Seville oranges or Seville orange-containing products, star fruit or star fruit-containing products within 7 days prior to dosing or intend to consume during the study
* Are unwilling to refrain from consuming xanthine-containing food and drink from 48 hours prior to admission until discharge from the CRU
* Have a defecation pattern less than once per day or acute constipation within 3 weeks prior to admission
* Have a history of clinically significant adverse drug reactions or "drug allergy" to more than 3 types of systemically administered medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3023414 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Baseline up to 144 hours postdose
Fecal Excretion of LY3023414 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Baseline up to 144 hours postdose

SECONDARY OUTCOMES:
Plasma Pharmacokinetics of LY3023414 and Radioactivity Maximum Observed Concentration (Cmax) | Baseline up to 144 hours postdose
Plasma Pharmacokinetics of LY3023414 and Radioactivity Time of Maximum Observed Concentration (Tmax) | Baseline up to 144 hours postdose
Plasma Pharmacokinetics of LY3023414 and Radioactivity Area Under the Concentration Versus Time Curve (AUC) | Baseline up to 144 hours postdose
Relative Abundance of LY3023414 and the Metabolites of LY3023414 as Measured by Percentage of Sample Radioactivity in Plasma, Feces, Urine | Baseline up to 144 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Madison, Wisconsin, United States